CLINICAL TRIAL: NCT01047982
Title: Myo-inositol May Prevent Gestational Diabetes in Obese Women
Brief Title: Myo-inositol in Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, associate professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INOGDM-2010
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; macrosomia; hypertension in pregnancy; HOMA-IR; obesity
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Obesity | interventions — Inositol; Folic Acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- myo-inositol (Active Comparator)
  Interventions: Dietary Supplement: myo-inositol
- placebo (Placebo Comparator): acid folic 400 mcg twice per day
  Interventions: Other: folic acid 400 mcg

INTERVENTIONS:
Dietary Supplement: myo-inositol — myo-inositol 2 grams plus folic acid 400 mcg twice a day
  Arms: myo-inositol
Other: folic acid 400 mcg — 2 pills a day
  Arms: placebo

SUMMARY:
Myo-Inositol is classified as a member of the vitamin B complex. It is a constituent of living cells and is widespread in many food. It is involved in a number of biological processes, including insulin signal transduction, resulting in modulating insulin sensitivity. This is a prospective, randomized, double center, placebo-controlled study. Two hundred and twenty obese pregnant women will be included in the trial and, after an informed consent, will assume randomly 2 g of myo-inositol twice a day or placebo from 12-13th weeks gestation until delivery. Then,they will perform an Oral Glucose Tolerance Test (OGTT) at 24-28th weeks gestation. Records about delivery (gestational age, neonatal weight...) will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Obese pregnant women: BMI > 30 Kg/cm2
* first trimester fast glycaemia < 126 mg/dl
* single pregnancy

Exclusion Criteria:

* Pregnant women with BMI < 30 Kg/cm2
* first trimester fast glycaemia > 126 mg/dl
* previous gestational diabetes
* twin pregnancy
* pregestational diabetes
* associated therapies with corticosteroids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
number of gestational diabetes cases diagnosed with OGTT | 24-28th weeks gestation
difference in HOMA values | from first trimester to OGTT

SECONDARY OUTCOMES:
incidence of pregnancy complications: hypertension, preterm delivery. macrosomia, shoulder dystocia, etc. | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, professor, Principal Investigator — University of Messina, ITALY
Locations (1):
- Obstetrics and Gynecology Unit, University of Messina and Obstetrics and Gynecology Unit of Modena University, Messina and Modena, Italy

REFERENCES:
- [Derived] Motuhifonua SK, Lin L, Alsweiler J, Crawford TJ, Crowther CA. Antenatal dietary supplementation with myo-inositol for preventing gestational diabetes. Cochrane Database Syst Rev. 2023 Feb 15;2(2):CD011507. doi: 10.1002/14651858.CD011507.pub3. PMID 36790138
- [Derived] D'Anna R, Di Benedetto A, Scilipoti A, Santamaria A, Interdonato ML, Petrella E, Neri I, Pintaudi B, Corrado F, Facchinetti F. Myo-inositol Supplementation for Prevention of Gestational Diabetes in Obese Pregnant Women: A Randomized Controlled Trial. Obstet Gynecol. 2015 Aug;126(2):310-315. doi: 10.1097/AOG.0000000000000958. PMID 26241420